CLINICAL TRIAL: NCT01213914
Title: The American Burn Association's Randomized Controlled Evaluation of Hemofiltration in Adult Burn Patients With Septic Shock and Acute Renal Failure
Brief Title: Hemofiltration in Burns: RESCUE (Randomized Controlled Evaluation of Hemofiltration in Adult Burn Patients With Septic Shock and Acute Renal Failure)
Acronym: RESCUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American Burn Association (Other)
Collaborators: United States Army Institute of Surgical Research (U.S. Federal Agency); Tampa General Hospital (Other); Medstar Health Research Institute (Other); Loyola University (Other); University of Texas Southwestern Medical Center (Other); Valleywise Health (Other); University of Tennessee (Other); University of Kansas Medical Center (Other); Doctors Hospital-Joseph M Still Burn Center (Unknown)
Responsible Party: Sponsor
Organization: United States Army Institute of Surgical Research (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-09-046; W81XWH-09-2-0194 (Other Grant/Funding Number: U.S. Army Medical Research and Materiel Command); Combat Casualty Grant (Other: American Burn Association)
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Burns; Hemofiltration; Kidney Failure, Acute; Shock, Septic
Keywords: Burns; Hemofiltration; Vasopressins; Kidney Failure Acute; Shock, Septic
MeSH Terms: conditions — Burns; Acute Kidney Injury; Shock, Septic; Diabetes Insipidus | interventions — Control Groups; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-volume hemofiltration at 70ml/kg/hr (Experimental): Paired randomization into four groups via central randomization center. Group 1: age 18-65 and <40%TBSA Group 2: age 18-65 and >40%TBSA Group 3: age >65 and <40%TBSA Group 4: age >65 and >40%TBSA
  Interventions: Device: An FDA approved continuous renal replacement device
- Control group (Active Comparator): Contemporary care via consideration of the Burn-Specific Sepsis Bundle adapted form the most recent Surviving Sepsis campaign recommendations and specifically modified to our patient population.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: An FDA approved continuous renal replacement device — 70ml/kg/hr for treatment group for 48 hours with the following requirements:
  * double lumen dialysis catheter should be placed in the internal jugular or femoral vein
  * Anticoagulation will be determined by prescribing physician
  * Use of 1.4 m2 or larger biocompatible synthetic hollow-fiber dialysis membrane that is changed every 24 hours
  * Blood flow rate will be set to ensure a filtration fraction of no more than 25%
  * Monitoring for electrolytes (specifically K+, Mg, Ca, and phos) during HVHF must be performed at least every 6 hours
  * Replacement fluids will be bicarbonate-buffered with appropriate adjustments when citrate-anticoagulation is utilized
  * All antibiotics will be dose adjusted for renal replacement therapy
  Other Names: High volume hemofiltration
  Arms: High-volume hemofiltration at 70ml/kg/hr
Other: Control Group — Both groups will receive 'contemporary' care via consideration of the Burn-specific Sepsis Bundle adapted from the most recent Surviving Sepsis Campaign (SSC) (1) recommendations and specifically modified to our patient population
  Other Names: Standard of care
  Arms: Control group

SUMMARY:
The purpose of this study is determine if High-Volume Hemofiltration in addition to 'contemporary' care will result in an improvement of select clinical outcomes when compared to 'contemporary' care alone in the treatment of critically ill patients with ARF secondary to septic shock.

DETAILED DESCRIPTION:
Acute renal failure (ARF) is a common and devastating complication in critically ill burn patients with mortality reported to be between 80 and 100%.(3-7) Despite recent advances in burn care, the unacceptably high mortality rate in this subgroup has not changed over time. The pathogenesis of ARF in burns, similar to other critically ill populations, is often multi-factorial with one major component being sepsis induced ischemic tubular necrosis. Thus, ARF secondary to septic shock is a common and devastating condition in the burn ICU.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the burn intensive care unit (ICU) with burns of any size
* Acute renal failure as previously defined by the Veterans Affairs/ National Institutes of Health (VA/NIH) Acute Renal Failure Trial Network study investigators(2)
* Patient is > 48 hours post-burn and in Septic Shock
* Patients 18 or older
* Patient/legally authorized representative willing to provide consent

Exclusion Criteria:

* Age <18
* Non-thermal injury (exfoliating skin disorders or necrotizing fasciitis)
* Pre-admission diagnosis of end stage renal failure
* Patients already on renal replacement therapy for more than 24 hours
* Patient not expected to survive more than 24 hours after randomization.
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-08; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Vasopressor dependency index | first 48 hours
  Vasopressor dependency index = MAP/Inotropic score • This index will correct for the inter-center variability that exists with regards to the point (minimum MAP) at which vasopressors are initiated or weaned off. Thus, this eliminates the need to 'standardize' starting/stopping criteria of vasopressors.
  Modified Inotropic index (30) = (dopamine dose X1)+(dobutamine dose X1)+(epi doseX100)+(norepi doseX100)+(phenylephrine doseX100)+(vasopressin doseX100)
  • All units recorded at each time point in mcg/kg/min
  Mean Arterial Pressure (mmHg)

SECONDARY OUTCOMES:
PaO2/FiO2 ratio and Oxygenation index | first 48 hours
Vasopressors-free days | first 14 days
Survival | 14 days, 28 days, and discharge
ICU days | Total number of days in ICU from date of Therapy Initiated through discharge
Ventilator free days | First 28 days after enrollment
Renal loss (need for long term renal replacement therapy) | greater than 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Kevin K Chung, MD, Study Chair — United States Army Institute of Surgical Research; Amy M Sprague, MD, Study Director — Doctors Hospital
Locations (9):
- United States (9):
  - Arizona Burn Center, Phoenix, Arizona
  - The Burn Center at Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Doctors Hospital-Joseph M Still Burn Center, Augusta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Regional Medical Center at Memphis, Memphis, Tennessee
  - University of Texas Southwestern Medical Center-Burn Center Parkland Health, Dallas, Texas
  - US Army Institute of Surgical Research, Fort Sam Houston, Texas

REFERENCES:
- [Background] VA/NIH Acute Renal Failure Trial Network; Palevsky PM, Zhang JH, O'Connor TZ, Chertow GM, Crowley ST, Choudhury D, Finkel K, Kellum JA, Paganini E, Schein RM, Smith MW, Swanson KM, Thompson BT, Vijayan A, Watnick S, Star RA, Peduzzi P. Intensity of renal support in critically ill patients with acute kidney injury. N Engl J Med. 2008 Jul 3;359(1):7-20. doi: 10.1056/NEJMoa0802639. Epub 2008 May 20. PMID 18492867
- [Background] Leblanc M, Thibeault Y, Querin S. Continuous haemofiltration and haemodiafiltration for acute renal failure in severely burned patients. Burns. 1997 Mar;23(2):160-5. doi: 10.1016/s0305-4179(96)00085-x. PMID 9177886
- [Background] Greenhalgh DG, Saffle JR, Holmes JH 4th, Gamelli RL, Palmieri TL, Horton JW, Tompkins RG, Traber DL, Mozingo DW, Deitch EA, Goodwin CW, Herndon DN, Gallagher JJ, Sanford AP, Jeng JC, Ahrenholz DH, Neely AN, O'Mara MS, Wolf SE, Purdue GF, Garner WL, Yowler CJ, Latenser BA; American Burn Association Consensus Conference on Burn Sepsis and Infection Group. American Burn Association consensus conference to define sepsis and infection in burns. J Burn Care Res. 2007 Nov-Dec;28(6):776-90. doi: 10.1097/BCR.0b013e3181599bc9. PMID 17925660
- [Background] Azevedo LC, Park M, Schettino GP. Novel potential therapies for septic shock. Shock. 2008 Oct;30 Suppl 1:60-6. doi: 10.1097/SHK.0b013e318181a425. PMID 18704007
- [Background] Ratanarat R, Permpikul C. Roles of extracorporeal blood purification in sepsis. J Med Assoc Thai. 2007 May;90(5):1021-31. PMID 17596062
- [Background] Chung KK, Lundy JB, Matson JR, Renz EM, White CE, King BT, Barillo DJ, Jones JA, Cancio LC, Blackbourne LH, Wolf SE. Continuous venovenous hemofiltration in severely burned patients with acute kidney injury: a cohort study. Crit Care. 2009;13(3):R62. doi: 10.1186/cc7801. Epub 2009 May 1. PMID 19409089
- [Background] Piccinni P, Dan M, Barbacini S, Carraro R, Lieta E, Marafon S, Zamperetti N, Brendolan A, D'Intini V, Tetta C, Bellomo R, Ronco C. Early isovolaemic haemofiltration in oliguric patients with septic shock. Intensive Care Med. 2006 Jan;32(1):80-6. doi: 10.1007/s00134-005-2815-x. Epub 2005 Nov 18. PMID 16328222
- [Background] Ronco C, Bellomo R, Homel P, Brendolan A, Dan M, Piccinni P, La Greca G. Effects of different doses in continuous veno-venous haemofiltration on outcomes of acute renal failure: a prospective randomised trial. Lancet. 2000 Jul 1;356(9223):26-30. doi: 10.1016/S0140-6736(00)02430-2. PMID 10892761
- [Background] Honore PM, Jamez J, Wauthier M, Lee PA, Dugernier T, Pirenne B, Hanique G, Matson JR. Prospective evaluation of short-term, high-volume isovolemic hemofiltration on the hemodynamic course and outcome in patients with intractable circulatory failure resulting from septic shock. Crit Care Med. 2000 Nov;28(11):3581-7. doi: 10.1097/00003246-200011000-00001. PMID 11098957
- [Background] Wagener G, Gubitosa G, Wang S, Borregaard N, Kim M, Lee HT. Urinary neutrophil gelatinase-associated lipocalin and acute kidney injury after cardiac surgery. Am J Kidney Dis. 2008 Sep;52(3):425-33. doi: 10.1053/j.ajkd.2008.05.018. Epub 2008 Jul 23. PMID 18649981
- [Background] Cruz DN, Antonelli M, Fumagalli R, Foltran F, Brienza N, Donati A, Malcangi V, Petrini F, Volta G, Bobbio Pallavicini FM, Rottoli F, Giunta F, Ronco C. Early use of polymyxin B hemoperfusion in abdominal septic shock: the EUPHAS randomized controlled trial. JAMA. 2009 Jun 17;301(23):2445-52. doi: 10.1001/jama.2009.856. PMID 19531784
- [Derived] Gibran NS, Shipper E, Phuong J, Braverman M, Bixby P, Price MA, Bulger EM; NTRAP Burns & Reconstructive Surgery Panel Group. Developing a national trauma research action plan: Results from the Burn Research Gap Delphi Survey. J Trauma Acute Care Surg. 2022 Jan 1;92(1):201-212. doi: 10.1097/TA.0000000000003409. PMID 34554139
- [Derived] Chung KK, Coates EC, Smith DJ Jr, Karlnoski RA, Hickerson WL, Arnold-Ross AL, Mosier MJ, Halerz M, Sprague AM, Mullins RF, Caruso DM, Albrecht M, Arnoldo BD, Burris AM, Taylor SL, Wolf SE; Randomized controlled Evaluation of high-volume hemofiltration in adult burn patients with Septic shoCk and acUte kidnEy injury (RESCUE) Investigators. High-volume hemofiltration in adult burn patients with septic shock and acute kidney injury: a multicenter randomized controlled trial. Crit Care. 2017 Nov 25;21(1):289. doi: 10.1186/s13054-017-1878-8. PMID 29178943